CLINICAL TRIAL: NCT01754272
Title: A Non-Interventional Follow-Up to the VELOUR Study (Multicentre International Study of Aflibercept Versus Placebo in Combination With FOLFIRI for Metastatic Colorectal Cancer) - Translational Research
Brief Title: A Non-Interventional Follow-Up to the VELOUR Study - Translational Research
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Sabine Tejpar, Professor, KU Leuven
Other Study IDs: ADX11080
Record Dates: First submitted 2012-12-12; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; mCRC; Aflibercept; FOLFIRI; translational research; retrospective; noninterventional; biomarkers; angiogenesis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived FFPE (Formaldehyde fixed paraffin-embedded) primary tumour colorectal cancer tissues Archived FFPE (Formaldehyde fixed paraffin-embedded) metastatic tumour tissue Archived residual blood samples (plasma, serum) collected in the frame of the VELOUR trial
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FOLFIRI + Aflibercept: Non-interventional study. No drugs administered. In this arm 612 patients from the VELOUR trial
- FOLFIRI + Placebo: Non-interventional study. 614 patients from the FOLFIRI + placebo arm in the VELOUR trial.

SUMMARY:
This is a follow-on study to the VELOUR trial (NCT00561470). The aim of this study is to acquire the archived colorectal cancer and metastasized tissue tumour blocks of patients who have participated in the VELOUR study.

These samples will be analysed to find proteins or markers which represent how an individual may be responding to treatment. The identification of these markers may help provide personalised and more effective treatment programs for patients with similar conditions in the future.

DETAILED DESCRIPTION:
The VELOUR trial (NCT00561470) has demonstrated the efficacy of aflibercept as a second line treatment in combination with fluorouracil, leucovorin, irinotecan (FOLFIRI)for metastatic colorectal cancer (mCRC) patients refractory to a first line oxaliplatin based chemotherapy regimen (Van Cutsem E., JCO 30 (2012):pp3499-3506). The FDA has approved Aflibercept (Zaltrap) for the treatment of metastatic colorectal cancer in combination with FOLFIRI on August 3rd 2012 and by European Medical Agency (EMEA) on November 15th 2012.

While the VELOUR study confirmed the benefits of using aflibercept in combination with FOLFIRI, the availability of biomarkers accurately predicting patients responding to this combination would further improve clinical utility of this drug. The molecular profiling of the Formaldehyde fixed paraffin embedded (FFPE) clinical tumor samples and serial plasma samples obtained from patients involved in VELOUR study and subsequent analysis of the molecular and clinical data would provide an invaluable opportunity to discover and potentially validate such biomarkers.

As blocks were not collected as part of the VELOUR trial, this protocol deals primarily with the steps that will be taken to gain ethics and consent in each of the participating countries and how the blocks will then be sourced and acquired, finally deposited in a biobank situated in KULeuven.

A VELOUR Translational Research Consortium (VTRC) has been formed by the Catholic University of Leuven (KULeuven)and Almac Diagnostics for the realisation of this study. The number of blocks available based on the surgical list held for the trial is estimated at 1030 (84% of complete trial cohort) and from a profiling viewpoint it has been calculated that the minimum number of blocks acceptable for processing and biomarker identification / validation is 500.

Due to the specific interest in angiogenesis, the VTRC consortium will aim to source blocks with both tumor and surrounding stromal tissue which will then be macro-dissected with the aim to generate data for both the tumor and surrounding angiogenic stroma. The project will generate gene expression, immunohistochemistry (IHC) and mutational data for these samples. In addition single nucleotide polymorphisms (SNP) data will be generated from non-tumor tissue, focusing on polymorphisms that demonstrate an association with disease or response outcome to therapy. Pre-processing and in silico evaluation of all data generated will support the outcome objectives of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have participated in the VELOUR trial

Exclusion Criteria:

* Patients who have not participated in the VELOUR trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastaic colorectal cancer who were refractory to an oxaliplatin-based chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1226 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Primary colorectal cancer tumor blocks | Two years
  Identify and acquire as many archived primary tumor blocks as possible of patients with mCRC treated in The VELOUR trial. Process the acquired samples as part of a translation research program.

SECONDARY OUTCOMES:
Metastatic tumor blocks | Two years
  Identify and acquire as many archived metastatic tumor tissue blocks as possible of patients with mCRC treated in The VELOUR trial. Process the acquired samples as part of a translation research program.Process the acquired samples as part of a translation research program

OTHER OUTCOMES:
Residual blood samples | Two years
  Acess as many residual blood samples (plasma, serum) collected in the frame of the VELOUR study as possible. Process the samples to determine markers relevant to angiogenesis factors, response to aflibercept and other markers which will be defined by the steering committee.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Tejpar, MD, PhD, Principal Investigator — KU Leuven
Locations (20):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia
- Medizinische Universität Wien, Vienna, Austria
- UZ Leuven UZ Gasthuisberg 3000 Leuven, Leuven, Belgium
- Hospital Sírio E Libanês, São Paulo, Brazil
- Odense Universitetshospital, Odense C, Denmark
- SA Põhja Eesti, Tartu, Estonia
- Universitaetsklinikum Halle (Saale), Halle, Germany
- University Hospital Of Heraklion Voutes, Heraklion, Crete, Greece
- IRCCS, Milan, Italy
- Orbis Medisch Centrum, Sittard-Geleen, Netherlands
- Oslo Universitetssykehus HF, Oslo, Norway
- Spitalul Universitar CF, Cluj-Napoca, Romania
- NN Blokhin Russian Cancer Research Center, Moscow, Russia
- Donald Gordon Medical Centre Wits University, Parktown, South Africa
- South Korea (2):
  - Samsung Medical Center Hematology and Oncology, Seoul
  - Asan Medical Center, Seoul
- Hospital Vall d'Hebrón, Barcelona, Spain
- Akademiska Sjukhuset Onkologiska Kliniken, Uppsala, Sweden
- Mount Vernon Hospital, Greater London, United Kingdom